CLINICAL TRIAL: NCT06488755
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Phase III Clinical Study Evaluating the Efficacy and Safety of SIM0718 in Adults and Adolescents With Asthma
Brief Title: SIM0718 Treatment of Asthma Clinical Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM0718-301
Record Dates: First submitted 2024-06-24; First posted 2024-07-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-06

CONDITIONS: Asthma; Eosinophilic
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: SIM0718 injection of placebo
- SIM0718 injection (Experimental): SIM0718 injection
  Interventions: Drug: SIM0718 injection

INTERVENTIONS:
Drug: SIM0718 injection — Dosage form: injection Specification: 300mg/2ml/bottle Dosage: A loading dose of 600 mg is injected subcutaneously on day 1, followed by 300 mg SIM0718 subcutaneously every two weeks.
  Duration of medication: 52 weeks
  Arms: SIM0718 injection
Drug: SIM0718 injection of placebo — Dosage form: injection Specification: 2ml/bottle Dosage: 4ml subcutaneously on day 1, followed by 2ml of placebo subcutaneously every two weeks.
  Duration of medication: 52 weeks
  Arms: Placebo

SUMMARY:
Phase III clinical study of SIM0718 asthma

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, parallel-group, placebo-controlled phase III clinical study evaluating the efficacy and safety of SIM0718 in adults and adolescents with asthma

ELIGIBILITY:
Inclusion Criteria:

* Age 12 to 75 years, weight ≥ 40 kg, diagnosed with asthma for at least 12 months；
* Currently receiving medium- to high-dose inhaled corticosteroids (ICS) in combination with 1 or 2 control medications and have been on a stable dose for at least 28 days prior to randomization；
* Pre-bronchodilator (trough) FEV1 ≤ 80% of predicted normal for adults and ≤90% of predicted normal for adolescents ；
* Positive bronchodilator response within 12 months prior to randomization or during the screening period;
* Asthma Control Questionnaire (ACQ-5) score ≥ 1.5;
* At least one severe asthma exacerbation within 12 months prior to the screening visit and no occurrence within 28 days prior to randomization;
* Based on the investigator judgment, the subject demonstrates acceptable inhaler, peak flow meter, and spirometry techniques;
* Compliance with usual asthma controller use ≥ 80% based on the patient diary in 7 days prior to dosing;
* Voluntarily participate in this clinical study and sign the informed consent form and be able to comply with the clinical visit schedule and study-related procedures;
* Female subjects of childbearing potential who are sexually active with non-sterilized male partners, male subjects, and their female partners of childbearing potential agree to use adequate and effective contraception throughout the study;

Exclusion Criteria:

* Current respiratory disease that may impair lung function as judged by the investigator;
* Diagnosis of helminth parasitic infection within 24 weeks prior to randomization and who have not received or have not responded to standard therapy;
* Within 28 days prior to randomization, with acute or chronic infection; or have a severe viral infection;
* Has a known or suspected history of immunosuppression or frequent, recurrent, or long-term infection;
* History of active tuberculosis; or untreated latent tuberculosis or tuberculosis not receiving standard treatment, unless the investigator judges that the patient has been adequately treated;
* People with hepatitis B, hepatitis C, or HIV infection;
* History of malignancy;
* Major surgery within 8 weeks prior to signing the informed;
* Bronchial thermoplasty within 12 months prior to randomization;
* Treatment of systemic glucocorticoid during 4 weeks prior to signing informed to randomization;
* Previous use or ongoing use of systemic immunosuppressants or biologics for the treatment of autoimmune or inflammatory diseases in 8 weeks or 5 half-lives prior to randomization;
* Within 16 weeks or 5 half-lives prior to randomization, received a biologic agent with the same therapeutic purpose;
* Participated in an interventional clinical trial of any drug or medical device within 3 months or 5 half-lives prior to randomization;
* Poor response to or intolerance to prior anti-IL-4Rα antibody therapy;
* Within 3 months prior to randomization, received specific immunotherapy；
* Receipt of intravenous human immunoglobulin (IVIG) or blood products within 30 days prior to randomization;
* Vaccination with live(attenuated) vaccine within 30 days prior to randomization or plan to receive live (attenuated) vaccine during the study;
* Are using concomitant medications or treatments that are prohibited in the protocol;
* The following laboratory abnormalities occurred during the screening period: eosinophils≥1500 cells/mm3 or 1.5×109/L; Platelets≤80,000 cells/mm3 or 80×109/L; phosphocreatine kinase (CPK) ≥5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) ≥3-fold ULN; aspartate aminotransferase (AST)≥ 3-fold ULN; Bilirubin ≥ 2x ULN;
* History of alcohol abuse or drug abuse within 12 months prior to randomization;
* Current smokers, or those who have been smoking in recent 6 months, or former smokers who have not been smoking for 6 months with a smoking history of ≥10 pack years;
* Allergy to L-histidine, trehalose, or Tween 80, or history of systemic hypersensitivity to any biologic products;
* Females of childbearing potential have a positive pregnancy test result during the screening period; Females planning to become pregnant or breastfeeding;
* Any clinically significant examination abnormality or serious and/or uncontrolled disease that, in the opinion of the investigator, may affect the subject safety, or affect the evaluation of efficacy, or preclude the subject completion of the entire study.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of severe asthma exacerbation events | 52 weeks
  Annualized rate of severe asthma exacerbation events within 52 weeks

SECONDARY OUTCOMES:
Change from baseline in forced expiratory volume in the first second before bronchodilator use | 12 weeks
  Change from baseline in forced expiratory volume in the first second before within 12 weeks
Change from baseline in Forced Vital Capacity (FVC) | During the 52-week treatment period
  Change from baseline in Forced Vital Capacity (FVC) of during the 52-week treatment period
Change from baseline in pre-bronchodilator forced expiratory volume in 1 second | During the 52-week treatment period
  Change from baseline in pre-bronchodilator forced expiratory volume in 1 second of during the 52-week treatment period
Change from baseline in Peak Expiratory Flow (PEF) | During the 52-week treatment period
  Change from baseline in Peak Expiratory Flow (PEF) of during the 52-week treatment period
Time from baseline to the first severe asthma exacerbation event, proportion of subjects with ≥ 1 severe asthma exacerbation | During the 52-week treatment period
  subjects with ≥ 1 severe asthma exacerbation of during the 52-week treatment period
Annualized rate of "loss of asthma control" events, time from baseline to "loss of asthma control"event | During the 52-week treatment period
  Annualized rate of "loss of asthma control" events, time from baseline to "loss of asthma control"event of during the 52-week treatment period
Change from baseline in annualized rate of hospitalization or emergency department visits, utilization of medical resources | During the 52-week treatment period
  Change from baseline in annualized rate of hospitalization or emergency department visits, utilization of medical resources of during the 52-week treatment period
Change from baseline in ASTHMA CONTROL QUESTIONNAIRE(ACQ-5) score | During the 52-week treatment period
  Change from baseline in ASTHMA CONTROL QUESTIONNAIRE(ACQ-5) score (5 questions, 0-6 score, higher score indicated lower asthma control) of during the 52-week treatment period
Asthma symptom score | During the 52-week treatment period
  Asthma symptom score (0-4 score, higher score indicated worse asthma symptom) during the 52-week treatment period
Use of rescue medication | During the 52-week treatment period
  Use of rescue medication of during the 52-week treatment period
Number of days of awakenings due to asthma and number of awakenings due to asthma | During the 52-week treatment period
  Number of days of awakenings due to asthma and number of awakenings due to asthma of during the 52-week treatment period
Change from baseline in standardized asthma quality of life questionnaire score ASTHMA QUALITY OF LIFE QUESTIONNAIRES(AQLQ(S)) | During the 52-week treatment period
  Change from baseline in standardized asthma quality of life questionnaire score(AQLQ(S)) (32 questions, 1-7 score, higher scores indicate better quality of life) of during the 52-week treatment period
Adverse events | during the 64 week study period
  Adverse events during 64 week study period
Vital signs | during the 64 week study period
  Vital signs during 64 week study period
Electrocardiograph (12-ECG) | during the 64 week study period
  Electrocardiograph (12-ECG) during 64 week study period
Laboratory tests | during the 64 week study period
  Laboratory tests during 64-week study period. Lab tests include hematology, biochemistry
SIM0718 blood concentration | During the 52-week treatment period
  SIM0718 blood concentration of during the 52-week treatment period
Positive rate and titer of anti-drug antibodies, positive rate of neutralizing antibodies | 64 weeks during the study
  Positive rate and titer of anti-drug antibodies, positive rate of neutralizing antibodies of 64 weeks during the study

CONTACTS AND LOCATIONS:
Overall Officials: L I hong zhuang, Study Director — Simcere Pharmaceutical Co., Ltd
Locations (1):
- China Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No